CLINICAL TRIAL: NCT04030130
Title: Parallel-Group, Randomized-Controlled Trial of Navigation Vs Usual Care for The Management of Delays and Racial Disparities Starting Adjuvant Therapy in Adults With Surgically-Managed, Locally Advanced HNSCC (NDURE 2.0)
Brief Title: Navigation vs Usual Care for Timely Adjuvant Therapy for Patients With Locally Advanced HNSCC
Acronym: NDURE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Evan Graboyes, Assistant Professor, Department of Otolaryngology-Head & Neck Surgery, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00091049-B; K08CA237858 (NIH)
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NDURE (Experimental): NDURE is a theory-based, multi-level patient navigation (PN) intervention consisting of three in-person, clinic-based sessions of manualized PN with multiple intervention components that target system-(care coordination), interpersonal-(social support), and individual- (health belief model [HBM]; perceived susceptibility, severity, barriers, self-efficacy) level health behavior theoretical constructs to reduce barriers to care, enhance HNSCC care delivery, and improve clinical outcomes (timely, equitable PORT). NDURE will be delivered from surgical consultation to PORT initiation (~3 months). The three in-person NDURE navigation sessions, which are expected to take 30-60 minutes each, will coincide with the presurgical consult, hospital discharge, and 1st postoperative clinic visit, time points chosen to facilitate case identification and coordination across key care transitions.
  Interventions: Behavioral: NDURE
- Usual Care (No Intervention): UC consists of discussions about the indications, risks/benefits/alternative, Guidelines, timing, and logistical details of adjuvant therapy. These discussions will be administered according to practice patterns of the involved providers.

INTERVENTIONS:
Behavioral: NDURE — NDURE is a theory-based, multi-level Patient Navigation (PN) intervention consisting of three in-person, clinic-based sessions of manualized PN with multiple intervention components that target system- (care coordination), interpersonal- (social support), and individual- (Health Belief Model; perceived susceptibility, severity, barriers, self-efficacy) level health behavior theoretical constructs to reduce barriers to care, improve cancer care delivery, and improve clinical outcomes (timely, equitable PORT). NDURE will be delivered from surgical consultation to PORT initiation (~3 months).
  Arms: NDURE

SUMMARY:
Head and neck cancer squamous cell carcinoma (HNSCC) is a disease with poor survival, especially for African Americans, despite intense treatment including surgery, radiation, and chemotherapy. Delays between surgery and the start of postoperative radiation therapy (PORT) are common, cause excess mortality, and contribute to worse survival in African Americans. Our research team has developed NDURE (Navigation for Disparities and Untimely Radiation thErapy), a novel theory-based patient navigation (PN) intervention to decrease delays and racial disparities starting PORT. In this single-site, open label, parallel-group, randomized controlled trial of adults with surgically-managed, locally advanced HNSCC, will be randomized to NDURE versus usual care to assess the preliminary clinical impact of NDURE on delays and racial disparities starting PORT after surgery for HNSCC. The investigators will collect information about the rate of PORT delay, racial disparities in the rate of PORT delay, and completion rate of key cancer care processes. Participants will also complete validated questionnaires at baseline and post-intervention to understand the theoretical constructs underlying NDURE . Post-intervention, patients and providers will undergo interviews to obtain in-depth understanding of the content, format, timing, and delivery of NDURE to optimize the intervention in preparation for a future multi-site study. NDURE could provide the first effective intervention to improve the delivery of timely, equitable PORT after HNC surgery, thereby improving survival for patients with HNC, decreasing racial disparities in mortality, and developing new standards of clinical care.

DETAILED DESCRIPTION:
Design: The study design is a Single-Site, Parallel-Group, Randomized-Controlled Trial of Navigation Versus Usual Care for The Management of Delays and Racial Disparities Starting Postoperative Radiation Therapy in Adults with Surgically-Managed, Locally Advanced Head and Neck Squamous Cell Carcinoma

Following screening and informed consent, sociodemographic, oncologic and symptom data will be prospectively gathered about participants from validated questionnaires and the electronic medical record (EMR). Participants will then be randomized to 3-sessions of the navigation intervention (NDURE; Navigation for Disparities and Untimely Radiation thErapy) or usual care (UC) and followed until the start of postoperative radiation therapy (PORT) following surgery for head and neck squamous cell carcinoma (HNSCC). Measures of PORT delay, racial disparities in PORT delay, key cancer care delivery processes, and theoretical constructs underlying PORT will be evaluated.

Treatment Allocation: Upon enrollment, participants will be randomized 1:1 to NDURE or UC using a stratified randomization design with strata defined by race (white, African American [AA]) and location of radiation facility (Medical University of South Carolina ([MUSC], non-MUSC) because of the known association of these variables with PORT delay.

Delivery of intervention:

NDURE is a theory-based, multi-level PN intervention consisting of three in-person, clinic-based sessions of manualized PN with multiple intervention components that target system- (care coordination), interpersonal- (social support), and individual- (Health Belief Model; perceived susceptibility, severity, barriers, self-efficacy) level health behavior theoretical constructs to reduce barriers to care, increase HNSCC care delivery, and improve clinical outcomes (timely, equitable PORT). NDURE will be delivered from surgical consultation to PORT initiation (~3 months). The NDURE intervention consists of: Navigation Sessions, the Navigator Manual, the Navigator Patient Guide, structured EMR documentation, weekly conferences to facilitate care coordination, real-time patient tracking, and multidisciplinary reporting. The three in-person NDURE navigation sessions, which are expected to take 30-60 minutes each, will coincide with the presurgical consult, hospital discharge, and 1st postoperative clinic visit, time points chosen to facilitate case identification and coordination across key care transitions. Contact beyond the three prescribed in-person sessions will occur with a frequency and modality (e.g. text message, email, etc.) dictated by patient and navigator need. During the first in-person session, the navigator will 1) elicit barriers and facilitators to timely PORT from the patient, caregiver, and provider, 2) develop the personalized barrier reduction plan (BRP), review it with the patient, caregiver, and provider, and 3) implement the BRP. At the two subsequent in-person sessions, the navigator will review and update the BRP in an iterative, dynamic fashion, identifying new barriers and systematically tracking resolution of prior barriers until the start of PORT. The Navigator Manual provides a structured resource to guide intervention delivery and enhance reproducibility. The Patient Guide is 1) literacy-level appropriate, 2) personalized for each patient's care pathway and BRP, 3) updated longitudinally as the patient progresses along the cancer continuum, and 4) available to patients in print and/or electronically via the patient portal in the EMR.

UC consists of oncology visits with provider-led discussion about the referrals needed to start PORT.

Expected Effect Size and Power Calculation: Power and sample size calculations were performed using PASS version 08.0.13, "Inequality Tests for Two Independent Proportions." The primary endpoint for this pilot RCT is the rate of PORT delay, defined by NCCN Guidelines as PORT initiation > 6 weeks following surgery. Our primary objective is to compare PORT delay rates between the NDURE and UC arms. Patients (n=150) will be randomized 1:1 to NDURE or UC using a stratified randomization design with strata defined by race (white or AA) and location of radiation facility (MUSC or not MUSC). Furthermore, to facilitate evaluation of PORT delay rates in racial subgroups, the investigators will oversample AAs for a final sample size of 50 white and 25 AA patients in each arm. The investigators assume the rate of PORT delay in the usual care arm will be 45% and target an absolute reduction of 20% for a PORT delay in the navigation arm of 25%. This effect size is clinically significant and is a realistic goal given published rates of improvement in similar (non-randomized) interventions. Seventy-five patients in each arm yields 83% power to detect a 20% reduction in PORT delay (45% versus 25%) based on a two-sided Mantel-Haenszel test of two independent proportions assuming a two-sided α = 0.1. Our choice of the Mantel-Haenszel test to compare proportions is based on the trial's stratified design. Our selection of α = 0.1 and 1 - β = 0.8 is based on the desire to emphasize power over type I error at this early stage of development (single institution phase II trial) to ensure follow-up on promising interventions. The investigators therefore consider our trial to be appropriately and rigorously designed to detect a clinically meaningful reduction in PORT delay.

Statistical Methods of Analysis: Graphical displays and descriptive statistics for sociodemographic, oncologic, and baseline symptom severity characteristics will be used to examine patterns and summarize data for each arm. The percentage of patients who start PORT within 6 weeks of surgery (the primary outcome measure) and corresponding 95% confidence interval (CI) will be calculated for both arms and for white and AA subgroups within each arm separately. The rate of PORT delay will be compared between arms using a Mantel-Haenszel test of two proportions, with strata defined by race and location of radiation facility. The investigators will analyze time to PORT as a continuous variable and estimate median time to PORT for each arm and for racial subgroups within each arm using Kaplan-Meier curves with Greenwood variance estimation to construct the corresponding 95% CIs. The investigators will estimate the hazard ratio comparing the two arms using Cox proportional hazards regression controlling for the stratification variables. The investigators will compare time to PORT between intervention arms using a stratified log-rank test. For other secondary endpoints, data will be summarized using frequency and percent for categorical variables and using mean, median, standard deviation, IQR and range for continuous variables. The investigators will also construct 95% CIs to provide a measure of uncertainty in estimated proportions and means. Comparisons between trial arms of other secondary endpoints will be performed using t-tests and chi-square tests, or Wilcoxon rank sum and Fisher's exact tests as appropriate. Baseline and post-intervention values of variables measuring the theoretical constructs underlying NDURE (i.e. care coordination, self-efficacy in cancer care, interpersonal support, and knowledge) will be compared using Wilcoxon sign rank tests. Comparisons between arms of the change in scores will be conducted using Wilcoxon rank sum tests.

ELIGIBILITY:
Inclusion Criteria:

Patient and disease characteristics

1. Age > 18 years at the time of screening
2. Histologically or pathologically confirmed invasive SCC (or histologic variant) of the oral cavity, oropharynx (p16 positive, negative, or unknown), hypopharynx, larynx, unknown primary, paranasal sinuses, or nasal cavity.

   a. In situations in which the patient fulfills all other inclusion criteria but the biopsy shows SCC in-situ or moderate/severe dysplasia (without definitive evidence of invasive SCC), but the patient is scheduled to undergo curative intent surgery by the treating oncologic surgeon due to clinical suspicion of invasive SCC, the diagnosis of SCC-in situ or moderate/severe dysplasia is sufficient to full the pathologic diagnosis enrollment criterion.
3. American Joint Committee on Cancer (AJCC) clinical stage grouping III-IV (8th edition) for patients with SCC of the oral cavity, p16-negative oropharynx, hypopharynx, larynx, paranasal sinuses, and nasal cavity; or AJCC clinical stage grouping III-IV (7th edition) for patients with p16-positive SCC of the oropharynx or unknown primary.

   1. At screening, AJCC clinical stage grouping should be determined based on a combination of physical exam, diagnostic evaluation with cross sectional imaging of the neck (computerized tomography (CT) and/or magnetic resonance imaging (MRI)) and/or 18-F-fluoro-deoxyglucose positron emission tomography (FDG PET) CT within 30 days
   2. In situations in which the patient fulfills all other inclusion criteria but the biopsy shows SCC in-situ or moderate/severe dysplasia (without definitive evidence of invasive SCC), but would otherwise have an appropriate clinical stage grouping as defined in criterion 5, the diagnosis of SCC-in situ or moderate/severe dysplasia is sufficient to full the staging enrollment criterion.
4. No prior exposure to radiation therapy, with or without concurrent chemotherapy, for treatment of HNSCC in the definitive or adjuvant therapy settings

   Surgery and adjuvant therapy eligibility
5. Plan for curative intent surgery at MUSC

   a. At screening, plan for curative intent surgical resection of the HNSCC at MUSC must be deemed likely by the treating surgeon and/or multidisciplinary tumor board, which must include a fellowship-trained head and neck oncologic surgeon
6. Plan for PORT (at MUSC or non-MUSC) with or without concurrent chemotherapy following curative intent surgery a. At screening, plan for adjuvant therapy following curative intent surgical resection of the HNSCC at MUSC must be deemed likely by the treating surgeon and/or multidisciplinary tumor board, which must include a fellowship-trained head and neck oncologic surgeon, based on the clinical expectation of at least one of the following adverse features on final pathologic evaluation: extranodal extension (ENE), pT3 or pT4 primary, N2 or N3 nodal disease, nodal disease in levels IV or V, perineural invasion (PNI), or lymphovascular invasion (LVI)

Exclusion Criteria:

1. Self-identified Hispanic ethnicity
2. Presence of cognitive impairment that precludes participation
3. Synchronous untreated malignancy
4. Failure to undergo curative intent surgery at MUSC
5. Lack of indication for PORT (with or without concurrent chemotherapy) per National Comprehensive Cancer Network (NCCN) Guidelines based on the presence of at least one of the following adverse features on final pathologic evaluation: ENE, positive margin, pT3 or pT4 primary, N2 or N3 nodal disease, nodal disease in levels IV or V, PNI, or LVI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graboyes EM, DeMass R, Sterba KR, Chera BS, Kistner-Griffin E, Hill EG, McCay J, Newman JG, Albergotti WG, Kejner AE, Skoner JM, Harper JL, Kaczmar J, Lee BJ, Zimmerman SA, Warren GW, Alberg AJ, Calhoun EA, Nussenbaum B, Hughes Halbert C. Randomized Trial of Enhanced Versus Standard Navigation to Promote Timely Initiation of Adjuvant Radiotherapy for Head and Neck Cancer. JCO Oncol Pract. 2025 Aug;21(8):1153-1164. doi: 10.1200/OP-24-00901. Epub 2025 Jan 6. PMID 39761486

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NDURE | Usual Care
Started | 88 | 88
Completed | 88 | 88
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NDURE | Usual Care | Total
Number analyzed (Participants) | 88 | 88 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 52 | 100
  >=65 years | 40 | 36 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (11.7) | 62.2 (10.8) | 62.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 27 | 61
  Male | 54 | 61 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 88 | 88 | 176
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 19 | 37
  White | 70 | 69 | 139
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 88 | 88 | 176
Predicted Location of PORT [Count of Participants; unit: Participants]
  MUSC | 27 | 25 | 52
  Not MUSC | 61 | 63 | 124

OUTCOME MEASURES:

1. Primary Outcome: Delay Initiating Postoperative Radiation Therapy (PORT)
Description: defined per National Comprehensive Cancer Network Guidelines as the initiation of PORT > 6 weeks (42 days) following definitive surgery for HNSCC
Time Frame: 6 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | NDURE | Usual Care
Number analyzed (Participants) | 67 | 78
Participants | 14 | 46

2. Secondary Outcome: Time Interval Between Surgery and the Start of PORT
Description: Time, in days, between the date of definitive surgical resection to the initiation of radiation therapy
Time Frame: 18 weeks from surgery
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | NDURE | Usual Care
Number analyzed (Participants) | 68 | 78
Days | 39 [36 to 40] | 47 [43 to 50]

3. Secondary Outcome: Treatment Package Time
Description: number of days from the date of definitive surgery for HNSCC to the date of PORT completion.
Time Frame: 18 weeks from surgery
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | NDURE | Usual Care
Number analyzed (Participants) | 64 | 71
Days | 84 [81 to 85] | 89 [87 to 94]

4. Secondary Outcome: Racial Differences in Delays in Starting PORT
Description: defined per National Comprehensive Cancer Network Guidelines as the initiation of PORT > 6 weeks (42 days) following definitive surgery for HNSCC between evaluable white and black patients with HNSCC
Time Frame: 6 weeks from surgery
Population: reporting PORT delay by racial subgroup
Measure: Count of Participants; unit: Participants
Arm/Group | NDURE | Usual Care
Number analyzed (Participants) | 67 | 78
Participants
  African American: number analyzed (Participants) | 11 | 19
  African American | 3 | 14
  White: number analyzed (Participants) | 56 | 59
  White | 11 | 32

5. Secondary Outcome: Racial Differences in Time Interval Between Surgery and the Start of PORT
Description: Difference between White and Black patients with HNSCC in the number of days between the date of definitive surgical resection to the initiation of radiation therapy.
Time Frame: 18 weeks from surgery
Population: reporting time to PORT by racial subgroup
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | NDURE | Usual Care
Number analyzed (Participants) | 68 | 78
Days
  African American: number analyzed (Participants) | 11 | 19
  African American | 38 [36 to 46] | 55 [43 to 60]
  White: number analyzed (Participants) | 57 | 59
  White | 39 [35 to 40] | 45 [42 to 49]

6. Secondary Outcome: Racial Differences in Treatment Package Time
Description: Difference between White and Black patients with HNSCC in the number of days from the date of definitive surgery for HNSCC to the date of PORT completion.
Time Frame: 18 weeks from surgery
Population: reporting racial differences in treatment package time
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | NDURE | Usual Care
Number analyzed (Participants) | 64 | 71
Days
  African American: number analyzed (Participants) | 10 | 17
  African American | 83 [78 to 89] | 93 [85 to 105]
  White: number analyzed (Participants) | 54 | 54
  White | 84 [81 to 85] | 88 [85 to 93]

7. Secondary Outcome: Percent of Patients With Pre-surgical Radiation Consultation
Description: The measures assesses the performance (or lack thereof) of a care delivery process (Pre-Surigcal Radiation Consultation) for patients with HNSCC. The measure is evaluated as performed if the patient attends a consultation with a radiation oncologist (at MUSC or elsewhere) prior to surgery to discuss RT in the definitive or adjuvant setting
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | NDURE | Usual Care
Number analyzed (Participants) | 68 | 78
Participants | 47 | 31

8. Secondary Outcome: Percent of Patients With Pre-Radiation Therapy Dental Extractions
Description: The measures assesses the performance (or lack thereof) of a care delivery process (Pre-Radiation Therapy Dental Extractions) for patients with HNSCC. The measure is evaluated as performed if the patient has extraction of his/her indicated teeth prior to discharge from the index hospitalization for the definitive surgical procedure. Patients who are edentulous are not evaluable for this measure.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | NDURE | Usual Care
Number analyzed (Participants) | 44 | 34
Participants | 44 | 31

9. Secondary Outcome: Time From Surgery to PORT Referral
Description: The measures assesses the time, in days, from the date of the definitive surgical procedure to the date the referral (or postoperative appointment) is placed to discuss adjuvant therapy with the treating radiation oncologist
Time Frame: 3 months
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | NDURE | Usual Care
Number analyzed (Participants) | 68 | 78
Days | 8 [8 to 9] | 16 [14 to 17]

10. Secondary Outcome: Time From Surgery to Postoperative Appointment With Radiation Oncology
Description: the time, in days, from the date of the definitive surgical procedure to the date that the patient attends a postoperative appointment with radiation oncology
Time Frame: 3 months
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | NDURE | Usual Care
Number analyzed (Participants) | 68 | 78
Days | 20.0 [19 to 21] | 24.5 [23 to 29]

ADVERSE EVENTS:
Time Frame: Recording/reporting of AEs will begin after the subject signs informed consent and end after the subject completes the intervention and follow up period as defined in the protocol. (18 weeks)
Description: N/a regarding differing definitions.
  This study did categorize AEs by severity and defined relationship to study for reporting.
Arm/Group | NDURE | Usual Care
All-Cause Mortality (participants affected / at risk) | 8/88 | 5/88
Serious Adverse Events (participants affected / at risk) | 0/88 | 0/88
Other Adverse Events (participants affected / at risk) | 0/88 | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT04030130/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT04030130/ICF_001.pdf